CLINICAL TRIAL: NCT04704622
Title: Comparative Evaluation of Intranasal Midazolam, Dexmedetomidine, Ketamine for Their Sedative Effect and the Ability to Facilitate Venous Cannulation in Pediatric Patients: a Prospective Randomized Study.
Brief Title: Comparison Between Dexmeditomidine, Midazolam and Ketamine as a Sedative to Help Cannula Insertion in Pediatric Patient
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rasha Gamal Abusinna, lecturer of anesthesia and intensive care, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Rasha Abusinna
Record Dates: First submitted 2021-01-04; First posted 2021-01-11 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Cannula Site Pain
Keywords: dexmedetomidine; ketamine; midazolam
MeSH Terms: interventions — Ketamine; TP63 protein, human; Midazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dexmedetomidine group (Active Comparator): dexmedetomidine intranasal injection,1 μg/kg, once, 30 min preoperative
  Interventions: Drug: Dexmedetomidine
- ketamine (Active Comparator): ketamine intranasal injection,2 mg/kg, once, 30 min preoperative
  Interventions: Drug: Ketamine
- midazolam (Active Comparator): midazolam intranasal injection,0.2 mg/kg, once, 30 min preoperative
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — ketamine intranasal injection,2 mg/kg, once, 30 min preoperative
  Other Names: ket
  Arms: ketamine
Drug: Midazolam — midazolam intranasal injection,0.2mg/kg, once, 30 min preoperative
  Other Names: mid
  Arms: midazolam
Drug: Dexmedetomidine — dexmedetomidine intranasal injection,1 μg/kg, once, 30 min preoperative
  Other Names: dex
  Arms: dexmedetomidine group

SUMMARY:
Background and Objectives: Surgery and hospitalization present a very stressful period for children and their parents. The induction of anesthesia and cannula insertion may be the only bad experience a child can remember during his procedure. Pediatric intravenous cannulation is technically difficult and moreover may cause psychological problems. Sedative Premedication has a great role in pediatric anesthesia to overcome fear and anxiety and to facilitate easy separation from their parents. Intranasal approach is safe and painless and well tolerated by children in addition to a comparable onset of action with the intravenous approach. Midazolam, dexmedetomidine and ketamine have proved their effectiveness as a sedative premedication. The objective of the current study was to compare the effectiveness of administration of intranasal midazolam, dexmedetomidine and ketamine as sedatives to facilitate and decrease the discomfort of intravenous cannulation before surgery in children undergoing various surgical procedures. Methods: the patients agreed to participate in the research were classified into 3 groups. Dexmedetomidine, Midazolam and Ketamine group; each group received the intranasal drug 30 min before the procedure. Pulse, MAP, oxygen saturation and sedation score (MOAA/S) baseline and every 10 min. Easiness of venipuncture, parental separation and any complication encountered were recorded.

DETAILED DESCRIPTION:
Background and Objectives: Surgery and hospitalization present a very stressful period for children and their parents. The induction of anesthesia and cannula insertion may be the only bad experience a child can remember during his procedure. Pediatric intravenous cannulation is technically difficult and moreover may cause psychological problems. Sedative Premedication has a great role in pediatric anesthesia to overcome fear and anxiety and to facilitate easy separation from their parents. Intranasal approach is safe and painless and well tolerated by children in addition to a comparable onset of action with the intravenous approach. Midazolam, dexmedetomidine and ketamine have proved their effectiveness as a sedative premedication. We assumed that intranasal midazolam, dexmedetomidine and ketamine would help anesthetics to carry out venous cannulation easily; in addition to their sedative premedication effect.

The objective of the current study was to compare the effectiveness of administration of intranasal midazolam, dexmedetomidine and ketamine as sedatives to facilitate and decrease the discomfort of intravenous cannulation before surgery in children undergoing various surgical procedures.

Study design: 150 patients agreed to participate in the research after written informed consent. patients were classified into 3 groups. Dexmedetomidine, Midazolam and Ketamine group; each group received the intranasal drug 30 min before the procedure. Pulse, MAP, oxygen saturation and sedation score (MOAA/S) baseline and every 10 min. Easiness of venipuncture, parental separation and any complication encountered were recorded. Group assignment, preparation and administration of drugs will be performed by a junior anesthetist who is neither involved nor interested by any means in the study.

ELIGIBILITY:
Inclusion Criteria: all the following must be included

* child aged between 2-9 years scheduled for minor elective surgical procedures (last 1-2 hours) at pediatric surgery department.
* Patients were ASA I or II.
* within normal range of weight.
* refusing venous cannulation

Exclusion Criteria: any of the following

* parents' refusal
* with nasal deformity or pathology
* any known case of allergy to the study drugs
* obese patients
* suspected difficult airway or venous cannulation.
* maxillofacial malformations
* gastroesophageal reflux
* patients with renal, liver, endocrine or cardiac pathology
* patients with increased intracranial or intraocular pressure
* patients with sleep apnea
* any patient with a preexisting cannula or accepting cannula insertion

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
the change of Modified Observer Assessment of Alertness and Sedation scale(MOAA/S) at different time intervals | measuring the Modified Observer Assessment of Alertness and Sedation scale every 10 minutes preoperative till induction of anesthesia up to 30 minutes
  scale measuring level of sedation from 1-6 points. 1 is referring to no sedation and 6 is the maximum sedation. reaching score of 4 is the sedation level needed to insert the cannula.

SECONDARY OUTCOMES:
the change in measuring pulse rate/ minutes at different time intervals | the recorded score at baseline and every 10 minutes preoperative till induction of anesthesia and intraoperative in a surgery 1-2 hours
  measuring pulse rate/ minutes every 10 minutes at baseline till the end of surgery
the change in Mean Arterial Pressure at different time intervals | the recorded score at baseline and every 10 minutes preoperative till induction of anesthesia and intraoperative in a surgery 1-2 hours
  measuring Mean Arterial Pressure every 10 minutes at baseline till the end of surgery
the change in oxygen saturation at different time intervals | the recorded score at baseline and every 10 minutes preoperative till induction of anesthesia and intraoperative in a surgery 1-2 hours
  measuring oxygen saturation every 10 minutes at baseline till the end of surgery
the ease of venipuncture score | done by the anesthetist immediately after the cannula insertion
  poor, fair, good, excellent

CONTACTS AND LOCATIONS:
Overall Officials: Rasha G Abusinna, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospital, Cairo, EL Abassia, Egypt

IPD SHARING:
Plan to Share IPD: No